CLINICAL TRIAL: NCT00049452
Title: A Randomized, Placebo Controlled Trial Of Zoledronic Acid For The Prevention Of Bone Loss In Premenopausal Women With Early Stage Breast Cancer
Brief Title: Zoledronate in Preventing Bone Loss in Premenopausal Women Receiving Chemotherapy After Surgery For Early Stage Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000258105; CPMC-IRB-14069; NCI-G02-2127; NOVARTIS-CPMC-IRB-14069
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
RATIONALE: It is not yet known whether zoledronate is effective in preventing bone loss in premenopausal women who are receiving adjuvant chemotherapy after undergoing surgery for early stage breast cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of zoledronate in preventing bone loss in premenopausal women who are receiving chemotherapy after surgery for early stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the changes in bone mineral density (BMD) and bone turnover that occur in premenopausal women with resected early stage breast cancer during and after 6 months of adjuvant chemotherapy.
* Determine the factors that predict bone loss during chemotherapy, particularly induction of amenorrhea, type of chemotherapeutic regimen, glucocorticoid exposure, and baseline BMD, in these patients.
* Determine whether zoledronate prevents bone loss in these patients when given during and after adjuvant chemotherapy.
* Determine the effect of zoledronate on markers of bone turnover in these patients during and after adjuvant chemotherapy.
* Determine whether the effect on markers of bone turnover predicts response to zoledronate in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to estrogen receptor status (positive vs negative), progesterone receptor status (positive vs negative), and adjuvant chemotherapy regimen. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive zoledronate IV over 15 minutes on day 1.
* Arm II: Patients receive placebo IV over 15 minutes on day 1. In both arms, treatment repeats every 3 months for up to 4 courses in the absence of disease progression. Patients also receive calcium and cholecalciferol (vitamin D) supplements daily.

Quality of life is assessed at baseline and at 6 and 12 months.

Patients are followed at 1 year.

PROJECTED ACCRUAL: A total of 120 patients (60 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized breast cancer

  * Stage I or II (T1-3, N0-2, M0)
* Planned adjuvant chemotherapy (after surgery) of at least 6 months in duration
* Hormone receptor status:

  * Estrogen receptor and progesterone receptor status known

PATIENT CHARACTERISTICS:

Age

* 18 to 50

Sex

* Female

Menopausal status

* Premenopausal or perimenopausal

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Creatinine less than 2 mg/dL

Other

* No T score of less than 2.0 on bone mineral density (BMD)
* No fragility fracture
* No lumbar spine anatomy that would preclude accurate BMD measurement of a minimum of 3 lumbar vertebrae
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 1 month since prior calcitonin
* At least 12 months since prior bisphosphonates given for more than 1 month duration
* No concurrent fluoride therapy (10 mg/day or more)
* No concurrent enrollment in another experimental drug study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2001-12; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Changes in lumbar spine bone mineral density (BMD) at 6 months

SECONDARY OUTCOMES:
Changes in lumbar spine BMD at 12 and 24 months
Total hip and femoral neck BMD at 6, 12, and 24 months
Serum markers of bone turnover (osteocalcin, bone-specific alkaline phosphatase, and cross-linked C-telopeptide of type 1 collagen levels) measured every 6 weeks for 6 months, and at 9 and 12 months
Quality of life as measured by the Short Form-36 instrument at baseline, and at 6 and 12 months
Treatment costs

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Carl and Dorothy Bennett Cancer Center at Stamford Hospital, Stamford, Connecticut
  - Valley Hospital - Paramus, Paramus, New Jersey
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York

REFERENCES:
- [Result] Hershman DL, McMahon DJ, Crew KD, Shao T, Cremers S, Brafman L, Awad D, Shane E. Prevention of bone loss by zoledronic acid in premenopausal women undergoing adjuvant chemotherapy persist up to one year following discontinuing treatment. J Clin Endocrinol Metab. 2010 Feb;95(2):559-66. doi: 10.1210/jc.2009-1366. Epub 2009 Dec 18. PMID 20022990
- [Result] Hershman DL, McMahon DJ, Crew KD, Cremers S, Irani D, Cucchiara G, Brafman L, Shane E. Zoledronic acid prevents bone loss in premenopausal women undergoing adjuvant chemotherapy for early-stage breast cancer. J Clin Oncol. 2008 Oct 10;26(29):4739-45. doi: 10.1200/JCO.2008.16.4707. Epub 2008 Aug 18. PMID 18711172
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716